CLINICAL TRIAL: NCT00161265
Title: UMCC 2004.064: Tissue Procurement Protocol for Patients Undergoing Neoadjuvant Systemic Therapy for Breast Cancer
Brief Title: Tissue Procurement Protocol for Patients Undergoing Neoadjuvant Systemic Therapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2004.064; IRB # 2005-009 and HUM 44194 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tissue and Organ Procurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: women with breast cancer
  Interventions: Procedure: tissue procurement

INTERVENTIONS:
Procedure: tissue procurement — tissue procurement

SUMMARY:
This study is being performed so that tumor and blood samples from patients who will receive breast cancer treatment prior to surgery can be collected and stored for future research.

DETAILED DESCRIPTION:
This protocol will provide a systematic approach to obtaining, cataloging, and distributing research tissue and blood from patients who will receive neoadjuvant systemic therapy for localized breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a primary measurable invasive breast cancer with the primary tumor intact (T1, 2, 3, or 4, any N, M0 or M1). Recurrent disease in the breast is also eligible.
2. The patient's clinical plan will include neoadjuvant systemic therapy (chemotherapy, hormonal therapy, biologic therapy), prior to surgery on the breast.
3. The clinical plan for patients with recurrent or M1 disease must include breast surgery after neoadjuvant systemic therapy. This would include patients with non-bulky M1 disease who the treating physicians feel would benefit from local control of disease after neoadjuvant systemic therapy.
4. Patients must have had mammography performed at the University of Michigan, OR outside film review prior to enrollment.
5. All patients are required to sign an informed consent regarding the experimental purpose of the research biopsies and serum banking, in accordance with the University of Michigan Institutional Review Board standards.

   -

Exclusion Criteria:

1. Breast tumors that are not measurable by any of the modalities, including physical examination, mammography, or ultrasound.
2. Tumors diagnosed by excisional biopsy, or incisional biopsy that does not leave measurable disease by physical examination, mammography, or ultrasound.
3. Patients must not have received any prior chemotherapy, hormonal therapy, or radiation therapy for their current breast cancer. Patients who received tamoxifen or other agents for prevention of breast cancer may be included.
4. Patients with another active systemic malignancy in the past year.

   -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2005-05; Primary Completion 2012-08 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne F. Schott, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided